CLINICAL TRIAL: NCT07337720
Title: Liposomal Amphotericin B in Patients With Invasive Aspergillosis and Hepatic Dysfunction: A Prospective Study
Brief Title: Liposomal Amphotericin B in Invasive Aspergillosis With Hepatic Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Principal Investigator, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZDSYLL264-P01
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Aspergillosis Invasive
Keywords: Invasive Aspergillosis; Liposomal Amphotericin B; Hepatic Dysfunction; Critically Ill Patients; Antifungal Therapy
MeSH Terms: conditions — Liver Diseases | interventions — liposomal amphotericin B; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-AmB group (Experimental): Patients with invasive aspergillosis complicated by hepatic dysfunction who are admitted to the intensive care unit (ICU) will be treated with liposomal amphotericin B (L-AmB) at a dose of 3 mg/kg/day administered by intravenous infusion for 2 weeks. Patients will then enter a 4-week follow-up period. During the follow-up period, investigators may decide to continue treatment with liposomal amphotericin B or switch to other antifungal agents based on the patients' clinical condition.
  Interventions: Drug: LIposomal amphotericin B (L-AmB) treatment

INTERVENTIONS:
Drug: LIposomal amphotericin B (L-AmB) treatment — Patients with invasive aspergillosis complicated by hepatic dysfunction who are admitted to the intensive care unit (ICU) will be treated with liposomal amphotericin B (L-AmB) at a dose of 3 mg/kg/day administered by intravenous infusion for 2 weeks. Patients will then enter a 4-week follow-up period. During the follow-up period, investigators may decide to continue treatment with liposomal amphotericin B or switch to other antifungal agents based on the patients' clinical condition.

SUMMARY:
Liposomal amphotericin B is an antifungal agent commonly used to treat invasive aspergillosis, a severe fungal infection associated with high mortality in critically ill patients. However, evidence regarding its safety and effectiveness in patients with hepatic dysfunction is limited.

In China, patients diagnosed with invasive aspergillosis complicated by hepatic dysfunction will be recruited from multiple centers. Eligible patients will receive treatment with liposomal amphotericin B according to the study protocol. The safety and effectiveness of liposomal amphotericin B in this patient population will be evaluated.

This study aims to provide clinical evidence to support antifungal treatment decisions for patients with invasive aspergillosis and impaired liver function.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, single-arm exploratory clinical study designed to evaluate the safety and effectiveness of liposomal amphotericin B (L-AmB) in critically ill patients with invasive aspergillosis complicated by hepatic dysfunction.

The study will be conducted in accordance with the principles of Good Clinical Practice and the Declaration of Helsinki. After approval by the ethics committees at all participating centers, eligible patients will be enrolled from 12 tertiary hospitals in China. Adult patients admitted to the intensive care unit (ICU) with a diagnosis of proven or probable invasive aspergillosis and concomitant hepatic dysfunction will be included according to predefined diagnostic and eligibility criteria.

All enrolled patients will receive liposomal amphotericin B as antifungal therapy at a dose of 3 mg/kg/day administered by intravenous infusion for a planned treatment duration of 2 weeks. Following completion of the initial treatment period, patients will enter a 4-week follow-up phase. During the follow-up period, investigators may decide to continue treatment with liposomal amphotericin B or switch to other antifungal agents based on the patients' clinical condition, liver function status, and current clinical practice guidelines.

Patients will be followed prospectively to assess treatment response, survival, and safety outcomes. The primary outcome of the study is overall response rate at Week 2 after initiation of liposomal amphotericin B therapy. Secondary outcomes include overall response rate at Week 6, survival rate at Week 6, clinical response, mycological response, changes in liver function parameters, incidence of adverse events and serious adverse events, length of intensive care unit stay, and overall survival.

This study aims to generate real-world clinical evidence on the use of liposomal amphotericin B in patients with invasive aspergillosis and hepatic dysfunction and to support optimized antifungal treatment strategies for this high-risk population in the intensive care setting.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following criteria to be eligible for enrollment:

1. Willing to participate in the study and able to provide written informed consent;
2. Hospitalized patients admitted to the intensive care unit (ICU);
3. Age ≥ 18 years, with no restriction on sex;
4. Proven or probable invasive aspergillosis (IA), defined as follows:

Proven IA

Proven IA is diagnosed if at least one of the following criteria is met:

1. Histopathological or cytopathological evidence of invasive Aspergillus spp. hyphae in tissue specimens obtained from a sterile site or the lung (e.g., biopsy or needle aspiration), with confirmation by culture or polymerase chain reaction (PCR);
2. Isolation of Aspergillus spp. by culture from a specimen obtained from a sterile site (e.g., biopsy or needle aspiration), with the lesion consistent with an infectious process.

Probable IA

Probable IA requires the presence of all of the following criteria:

1. At least one host factor (e.g., COVID-19, influenza, solid malignancy, HIV infection with CD4 <200 cells/µL, decompensated liver cirrhosis, or moderate to severe chronic obstructive pulmonary disease [COPD]);
2. At least one compatible clinical feature (e.g., fever ≥38.3 °C lasting ≥3 days, pleuritic chest pain, dyspnea, hemoptysis, or worsening respiratory failure despite appropriate antibacterial therapy);
3. At least one compatible radiological finding (e.g., newly developed pulmonary infiltrates on chest computed tomography, or cavitary lesions not explained by other causes);
4. At least one mycological criterion (e.g., positive culture for Aspergillus spp. from bronchoalveolar lavage fluid [BALF], serum galactomannan >0.5 optical density index [ODI], or BALF galactomannan ≥1.0 ODI).
5. Concomitant hepatic dysfunction meeting at least one of the following conditions:

   * Aminotransferase levels >3 times the upper limit of normal (ULN) and <10 times ULN;
   * Child-Pugh class A or B;
6. Expected to receive antifungal therapy for ≥5 days.

Exclusion Criteria

Patients meeting any of the following criteria will be excluded:

1. Pregnant or breastfeeding women;
2. Known allergy or hypersensitivity to amphotericin B or any of its formulations;
3. Previous treatment with extracorporeal membrane oxygenation (ECMO);
4. Expected life expectancy <48 hours;
5. Patients who, at the time of enrollment, are confirmed to require antifungal agents other than those specified in the study protocol;
6. Presence of any of the following severe comorbid conditions that may interfere with assessment of study efficacy or safety:

   * Acute liver failure or acute decompensation of chronic liver failure;
   * Known or suspected active pulmonary tuberculosis, cystic fibrosis, lung abscess, empyema, or obstructive pneumonia;
7. Severe renal impairment, defined as any of the following:

   * Creatinine clearance (CrCL) <16 mL/min at enrollment;
   * Requirement for hemodialysis, peritoneal dialysis, or other renal replacement therapy at enrollment;
8. Participation in another clinical trial within 3 months prior to enrollment;
9. Previous enrollment in this study;
10. Any condition that may affect study compliance or outcome assessment (e.g., planned major surgery, or inability to comply with the study protocol due to disease severity or poor adherence);
11. Any other condition deemed by the investigator to make the patient unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
2 weeks Overall response rate | from treatment begin to Week 2
  Overall response rate

SECONDARY OUTCOMES:
6 weeks Overall response rate | from treatment begin to week 6
  Overall response rate
6 weeks Survival rate | from treatment begin to week 6
  Survival rate

IPD SHARING:
Plan to Share IPD: No